CLINICAL TRIAL: NCT01063257
Title: A Phase I/II Multicenter Study of IV Clofarabine in Patients With High-Risk Myelodysplastic Syndrome Who Have Failed Therapy With Azacitidine: the NIDEVOL Study
Brief Title: Clofarabine in High Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFM-CLO-08
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A (Experimental): Clofarabine treatment at D1-D5
  Interventions: Drug: Clofarabine
- Cohort B (Experimental): Clofarabine treatment at D1, D3, D5, D8, D10
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — The dosage of Clofarabine will be gradually augmented in a 3+3 design for each following dose level:
  DL1 - 5mg/m2/d, DL2 - 7.5mg/m2/d, DL3 - 10mg/m2/d, DL4 - 12.5mg/m2/d (This dose may not be reached and is an optional dose level in case the MTD is not reached before and depending on further data from the ongoing MDS Phase IIa oral formulation trial).
  The DLa will be the following:
  DL1a - 2.5mg/m2/d, DL2a - 6.5mg/m2/d, DL3a - 8.5mg/m2/d, DL4a - 11.5mg/m2/d (In case of activation of the DL4 step). Dose levels 1a, 2a and 3a will be used for de-escalation.
  Other Names: EVOLTRA®

SUMMARY:
This study aims to determine the maximal tolerated dose (MTD) and dose limiting toxicities (DLTs) of low dose IV clofarabine for MDS patients after treatment failure of azacitidine.

DETAILED DESCRIPTION:
The study is an open-label, 3+3 dose-escalation, phase I/II study.The duration of enrollment in the phase I study is 12 months.

Fourteen patients will be enrolled at the RD using the selected dosing in each cohort, for an enrollment period of 12 months.

Each patient may receive up to 8 courses, every 4 to 8 weeks in a D1-D5 schedule or every other day from D1 to D10.

Each patient will be followed for up to 24 months.

Primary endpoint of the phase I part:

* To determine the maximal tolerated dose (MTD) and dose limiting toxicities (DLTs) of increased doses of IV clofarabine administered either daily from D1 to D5 for a 28 to 56 day-course or every other day from D1 to D10 for a 28 to 56 day-course.

Secondary endpoints:

* To determine response rates, as defined by the 2006 modified IWG criteria, associated with the two different dosing and scheduling of clofarabine in patients with high-risk MDS or AML patients with less than 30% marrow blasts (RAEB-T in FAB MDS classification), previously treated by azacitidine and without erythroid response after 6 cycles of azacitidine.
* To evaluate response duration, time to IPSS progression, and loss of RBC transfusion independence in these patients.
* To evaluate hospitalization duration, rates of rehospitalization for non-hematological toxicities, severe bleeding or febrile neutropenia.

If treatment is feasible the study will be extended to the phase II part.

Study Objectives:

Primary endpoint:

* To confirm safety and hematological toxicity in 14 additional patients. Secondary endpoints
* To evaluate response duration, time to IPSS progression, and loss of RBC transfusion independence in these patients.
* To evaluate hospitalization duration, rates of rehospitalization for non hematological toxicities, severe bleeding or febrile neutropenia.
* To determine the response rate as defined by the 2006 modified IWG criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more with MDS according to FAB classification and intermediate-2 or high IPSS risk scores, or CMML (with WBC < 13 x 109/L and bone marrow blasts > 10 %) according to WHO classification, or AML according to WHO classification if less than 30 % bone marrow blasts (RAEB-T according to FAB MDS classification or AML according to WHO classification with more than 30 % with bone marrow blasts only if preceded by a proven MDS phase.
* Patients previously treated by azacitidine (Vidaza®) in proven progression, or stable after 6 courses with ongoing transfusion dependent anemia (> 4 RBC units in the 8 weeks preceding inclusion (as erythroid response in IWG 2006 criteria is reduction of at least 4 RBC units in 8 weeks).
* Previous biological and or targeted therapies of MDS or AML are allowed if stopped more than 1 month before inclusion.
* ECOG PS ≤ 2.
* Adequate renal and liver function :

  i.e. Serum creatinine < 110 microM in men or 90 microM in women. If plasma creatinine level < 90 - 110 microM, then the estimated glomerular filtration rate (GFR) must be < 50 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease (MDRD) equation where Predicted GFR (mL/min/1.73 m2) = 32788 x (plasma creatinine level (microM)-1.154 x (age in years)-0.023 x (0.742 if patient is female) x (1.212 if patient is African American)
* Bilirubin < 1.5 x ULN, (except increased unconjugated bilirubin due to dyserythropoiesis).
* Aspartate transaminase (AST)/alanine transaminase (ALT) < 2.5 × ULN and Alkaline phosphatase < 2.5 × ULN.
* Absence of pregnancy or lactation in female patients (Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment).
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.
* Provided signed written informed consent.
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.

Exclusion Criteria:

* Patients with AML and bone marrow blasts count of 20-30%, if candidates to intensive AML type chemotherapy.
* Known hypersensitivity to clofarabine or excipients.
* Concomitant malignant disease.
* Active uncontrolled infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Concomitant severe cardiovascular disease, i.e. congestive heart failure (NYHA grade > 3).
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* No affiliation to a national insurance scheme directly or to an equivalent system.
* Chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
* Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea. The patient must have recovered from all acute toxicities from any previous therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To determine the maximal tolerated dose (MTD) and dose limiting toxicities (DLTs) | 1-2 months
  After one course treatment.

SECONDARY OUTCOMES:
To determine response rates. | 1-16 months.
  After one, two and eight courses of treatment.
To evaluate the response duration. | 1-16 months
  After one, two and eight courses of treatment.
To evaluate time to IPSS progression. | 1-16 months
  After one, two and eight courses of treatment.
To evaluate loss of RBC transfusion independence and hospitalization duration. | 1-16 months
  After one, two and eight courses of treatment.
To evaluate rates of rehospitalization for non-hematological toxicities, severe bleeding or febrile neutropenia. | 1-16 months
  After one, two and eight courses of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Braun, MD, Principal Investigator — Groupe Francophone des Myélodysplasies; Claude Gardin, MD, Study Chair — Groupe Francophone des Myélodysplasies
Locations (5):
- France (5):
  - Hôpital Avicenne, Bobigny
  - Institut Paoli-Calmettes, Marseille
  - Hôpital Saint-Louis, Paris
  - Hopital Cochin Service d'Hématologie, Paris
  - Centre Henri Becquerel, Rouen

REFERENCES:
- See also: Website of the Groupe Francophone des Myélodysplasies (GFM) — http://www.gfmgroup.org